CLINICAL TRIAL: NCT07005778
Title: Effects of Traditional Pain Education and Pain Neuroscience Education on Pain Attitudes and Beliefs in Physiotherapy Assistant Students
Brief Title: Effects of Pain Neuroscience Education on Pain Attitudes and Beliefs in Physiotherapy Assistant Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hatice Gül, Head of Therapy and Rehabilitation Department of Vocational School of Health Services, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 03.10.2024, TBAEK-683
Record Dates: First submitted 2025-05-26; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Pain Education (Active Comparator): Participants in the control group received a 70-minute lecture based on the biomedical model of pain.
  Interventions: Other: Traditional pain education
- PNE based education (Experimental): Students in the intervention group received a 70-minute lecture grounded in the biopsychosocial model of pain.
  Interventions: Other: PNE-based education

INTERVENTIONS:
Other: Traditional pain education — Participants in the control group received a 70-minute lecture based on the biomedical model of pain. Educational content included anatomical pathways for pain process (receptors, Aδ and C fibers, spinal cord, and ascending tracts), mechanisms of action potential generation, and the Gate Control Theory. The role of the brain was briefly addressed in the context of descending inhibition. While the Neuromatrix Theory was mentioned, the presentation lacked metaphorical or narrative-based content. Case examples centered on inflammation and tissue injury.
  Arms: Traditional Pain Education
Other: PNE-based education — Students in the intervention group received a 70-minute lecture grounded in the biopsychosocial model of pain. The session emphasized that pain is not a direct result of tissue damage, but rather a complex and context-dependent output of the brain. The lecture explored how pain emerges from the brain's interpretation of various inputs, including sensory signals, prior experiences, beliefs, emotions, and environmental factors.
  Instructional strategies included the use of clinically relevant metaphors and storytelling to promote reconceptualization of pain. Examples such as "the alarm system" were used to illustrate peripheral and central sensitization, while real-life anecdotes (a player unaware of injury during a game or a nail-in-foot case with no significant damage) highlighted the dissociation between nociception and pain experience.
  Arms: PNE based education

SUMMARY:
The goal of this educational trial is to learn whether Pain Neuroscience Education (PNE) improves pain-related attitudes and beliefs in physiotherapy assistant (PTA) students in Turkey compared to traditional pain education. The main questions this study aims to answer are:

Does a single-session PNE-based education improve students' beliefs about the relationship between pain and disability? Does it reduce reliance on biomedical (organic) pain beliefs compared to traditional pain education? In this study, researchers will compare PNE-based education to traditional pain education, both delivered through 70-minute lectures.

Participants were randomly assigned to either the PNE group or the traditional education group, attended a one time 70-minute classroom lecture, completed questionnaires at three time points: before the session, immediately after, and 3 months later.

The main tools used will be the Health Care Providers' Pain Attitudes and Impairment Relationship Scale (HC-PAIRS) and the Pain Beliefs Questionnaire (PBQ), which includes organic and psychological subscales.

This study aims to support the integration of contemporary pain neuroscience content into physiotherapy assistant curricula to enhance biopsychosocial understanding at an early stage of professional education.

DETAILED DESCRIPTION:
In Turkey, research on the impact of pain neuroscience education (PNE) on the knowledge, beliefs, and attitudes of undergraduate physiotherapy students remains scarce. Moreover, there appears to be no study that directly contrasts traditional pain education with a PNE-based approach that conceptualizes pain as an outcome-driven process, enriched with metaphors and storytelling. Existing literature suggests that physiotherapy assistant programs often provide limited exposure to neuroscience content, which may contribute to the lack of significant improvements in students' understanding and attitudes toward pain following PNE.

Against this background, the current study was developed to explore how a metaphor-supported, case-based PNE intervention influences the pain-related knowledge and beliefs of physiotherapy assistant students. To the best of our knowledge, no prior study in Turkey has systematically evaluated the effects of PNE within this specific student group. Therefore, a randomized controlled trial was designed to compare the outcomes of traditional structural pain education and a neuroscience-based educational program on pain-related beliefs and attitudes among physiotherapy assistant students.

ELIGIBILITY:
Inclusion Criteria:

* Students were eligible to participate if they were undergraduate physiotherapy assistant students enrolled at the Vocational School of Health Services.

Exclusion Criteria:

* Individuals were excluded if they had previously received in-depth teaching on pain neurophysiology or traditional pain education.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
The Health Care Pain Attitudes and Impairment Relationship Scale | Participants completed the HC-PAIRS at baseline, Day 1 and 3 months.
  The HC-PAIRS is a 12-item scale that measures healthcare providers' beliefs about how much pain leads to disability in low back pain cases, using a 7-point Likert scale. Higher scores indicate more negative attitudes. The Turkish version was validated and showed strong reliability (ICC = 0.85).

SECONDARY OUTCOMES:
Pain Beliefs Questionnaire | Participants completed the Pain Beliefs Questionnaire at baseline, Day 1 and 3 months
  The Pain Beliefs Questionnaire (PBQ) is a 12-item tool designed to assess individuals' beliefs about pain, divided into two subscales: Organic (8 items) and Psychological (4 items). The Organic subscale reflects beliefs about the physical causes of pain, while the Psychological subscale focuses on the influence of emotional and mental states such as anxiety and relaxation. Items are rated on a 6-point scale ranging from "always" to "never." Subscale scores are calculated by summing the relevant items. The PBQ can be used with healthy individuals and has been shown to have valid and reliable psychometric properties in its Turkish version.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Gül, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the dataset includes personal data, it is not planned to be shared.

REFERENCES:
- [Result] Mankelow J, Ryan C, Taylor P, Martin D. The effect of pain neurophysiology education on healthcare students' knowledge, attitudes and behaviours towards pain: A mixed-methods randomised controlled trial. Musculoskelet Sci Pract. 2020 Dec;50:102249. doi: 10.1016/j.msksp.2020.102249. Epub 2020 Aug 28. PMID 32920228
- [Result] Cox T, Louw A, Puentedura EJ. An abbreviated therapeutic neuroscience education session improves pain knowledge in first-year physical therapy students but does not change attitudes or beliefs. J Man Manip Ther. 2017 Feb;25(1):11-21. doi: 10.1080/10669817.2015.1122308. Epub 2016 Feb 10. PMID 28855788
- [Result] Colleary G, O'Sullivan K, Griffin D, Ryan CG, Martin DJ. Effect of pain neurophysiology education on physiotherapy students' understanding of chronic pain, clinical recommendations and attitudes towards people with chronic pain: a randomised controlled trial. Physiotherapy. 2017 Dec;103(4):423-429. doi: 10.1016/j.physio.2017.01.006. Epub 2017 Mar 22. PMID 28797666